CLINICAL TRIAL: NCT04083937
Title: Prostate Cancer Patients Treated With Alternative Radiation Oncology Strategies
Acronym: PAROS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAROS
Record Dates: First submitted 2019-01-07; First posted 2019-09-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Photons; Protons

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 70.0/ 2.0 Gray (RBE) (Active Comparator): Normofractionated radiotherapy with photons (70.0/ 2.0 Gray)
  Interventions: Radiation: Normofractionated radiotherapy with photons
- 57.0/ 3.0 Gray (RBE) (Experimental): Hypofractionated radiotherapy with photons (57.0/ 3.0 Gray)
  Interventions: Radiation: Hypofractionated radiotherapy with photons
- 57.0/ 3.0 (RBE) (Experimental): Hypofractionated radiotherapy with protons (57.0/ 3.0 Gray relative biological effectiveness [RBE]).
  Interventions: Radiation: Hypofractionated radiotherapy with protons

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy with photons — hypofractionated radiotherapy with photons (total dose 57.0 Gray in 19 fractions)
  Arms: 57.0/ 3.0 Gray (RBE)
Radiation: Hypofractionated radiotherapy with protons — hypofractionated radiotherapy with protons (total dose 57.0 Gray relative biological effectiveness (RBE) in 19 fractions)
  Arms: 57.0/ 3.0 (RBE)
Radiation: Normofractionated radiotherapy with photons — normofractionated radiotherapy with photons (total dose 70.0 Gray in 35 fractions)
  Arms: 70.0/ 2.0 Gray (RBE)

SUMMARY:
As the most common male carcinoma, prostate cancer is a major tumor entity in oncology. In addition to definitive radiotherapy, surgical procedure is considered to be an oncologically equivalent therapeutic alternative for non-metastatic malignancies in the primary setting. However, a subsequent radiotherapy of the prostate bed is often necessary, which takes place as an "adjuvant" treatment immediately after surgery or in the course of a repeated increase in PSA and usually extends over several weeks. For the primary situation (without previous surgery), several randomized phase III clinical trials have shown that it is possible to shorten radiotherapy by increasing the single dose (called hypofractionation). In the context of two prospective Phase II studies, which were carried out in Heidelberg, it has since been shown that hypofractionation with both photons and protons is safe and feasible even in the postoperative situation.

The current, prospective and randomized PAROS study is now intended to demonstrate a multicentric phase III study as an improvement in the quality of life caused by rectum toxicity (primary endpoint) by the use of protons. The oncological non-inferiority of hypofractionated radiotherapy after surgery is a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* histology-proven prostate cancer with Gleason Score and PSA-value;
* indication for prostate bed irradiation (adjuvant/ salvage) after prostatectomy;
* Karnofsky-Index ≥ 70%
* age ≥ 18 years

Exclusion Criteria:

* androgen deprivation therapy
* lymphatic spread
* macroscopic tumor/ R2
* stage IV (M1)
* previous irradiation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 897 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (prostate-associated, 12 weeks vs baseline) | 12 weeks
  The primary objective of the present trial is to show a Change in the bowel symptoms according to scores on the EORTC QLQ-PR25 questionaire after proton therapy compared to photon irradiation (week 12 vs. baseline).

SECONDARY OUTCOMES:
biochemical progression-free survival (bPFS) | 5 years after baseline
  non-inferiority of hypofractionated radiotherapy compared to normofractionated radiotherapy with regard to biochemical progression-free survival (bPFS)
overall survival (OS) | 5 years after baseline
  non-inferiority of hypofractionated radiotherapy compared to normofractionated radiotherapy with regard to overall survival (OS)
Toxicity acc. to NCI CTCAE V 5.0 after 2 and 5 years | 2 and 5 years after baseline
  non-inferiority of hypofractionated radiotherapy compared to normofractionated radiotherapy with regard to toxicity
Quality of life (general and prostate-associated, 2 years and 5 years vs. baseline) | 2 and 5 years after baseline
  non-inferiority of hypofractionated radiotherapy compared to normofractionated radiotherapy with regard to changes in the scores of quality of life based on the EORTC QLQ-C30 questionaire
Quality of life (general and prostate-associated, 2 years and 5 years vs. baseline) | 2 and 5 years after baseline
  non-inferiority of hypofractionated radiotherapy compared to normofractionated radiotherapy with regard to changes in the scores of quality of life based on the EORTC QLQ-PR25 questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany